CLINICAL TRIAL: NCT05416606
Title: Transurethral Bipolar Enucleation and Resection of the Prostate Versus Open Prostatectomy for the Treatment of Benign Prostatic Hyperplasia
Brief Title: Prostate Bipolar Enucleation and Resection Versus Open Prostatectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helwan University (Other)
Responsible Party: Principal Investigator, Mohamed Fawzy Hassan Mahdy Elsyaad, Principal Investigator, Helwan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 51-2020
Record Dates: First submitted 2022-06-05; First posted 2022-06-13 (Actual); Last update posted 2022-06-13 (Actual); Status verified 2022-06

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: Transurethral enucleation; Transurethral enucleation and resection of the prostate; plasma enucleation; prostate enucleation; Open Prostatectomy; BPH; Benign prostatic hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Prostatectomy

STUDY DESIGN:
Intervention Model Description: In this study, a hybrid technique, that combines two types of techniques using the same cutting current and technological setup, will be proposed enucleation of the prostate gland with the plasma vaporization electrode and resection with a TURis cutting loop. This technique is defined as transurethral vapor enucleation and resection of the prostate (TVERP) comparing it with open prostatectomy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- transurethral bipolar enucleation and resection of the prostate (Active Comparator): transurethral bipolar enucleation and resection of the prostate
  Interventions: Procedure: transurethral bipolar enucleation and resection of the prostate
- open prostatectomy (Active Comparator): open surgical transvesical prostatectomy
  Interventions: Procedure: open surgical transvesical prostatectomy

INTERVENTIONS:
Procedure: transurethral bipolar enucleation and resection of the prostate — transurethral bipolar enucleation and resection of the prostate
  Other Names: TUVERP
  Arms: transurethral bipolar enucleation and resection of the prostate
Procedure: open surgical transvesical prostatectomy — open surgical transvesical prostatectomy
  Other Names: Transvesical prostatectomy
  Arms: open prostatectomy

SUMMARY:
Benign prostatic hyperplasia (BPH) is a frequent disease in aging men accompanied by bladder outlet obstruction (BOO). Open prostatectomy (OP) is still considered the first-line treatment for more than 80 ml prostate size. In this study, a mixed technique called transurethral bipolar enucleation and resection of the prostate (TBERP) was compared to the standard open prostatectomy.

DETAILED DESCRIPTION:
Benign prostatic hyperplasia (BPH) is a frequent disease in aging men accompanied by bladder outlet obstruction (BOO). Open prostatectomy (OP) is still considered the first-line treatment for more than 80 ml prostate size. In this study, a mixed technique called transurethral bipolar enucleation and resection of the prostate (TBERP) was compared to the standard open prostatectomy.

This is a Comparative, Prospective Study conducted on men over 50 years.The patients were randomly distributed into two groups treated by TBERP and OP. Patients were evaluated preoperatively and at 1-week post catheter removal and 1-3-months postoperatively in terms of blood loss, operation time, the weight of resected prostatic tissues, post-operative catheterisation period, hospital stay, IPSS, PVR, prostate volume, early complications (recatheterization, urine retention, UTI and irritative symptoms) and late complications (urinary incontinence, urethral stricture and bladder neck contracture).

ELIGIBILITY:
Inclusion Criteria:

* Male patients
* Age more than 50 years
* Prostate size of more than 80 ml
* IPSS ≥ 8, and maximum urinary flow rate (Qmax) ≤ 15 mL/s
* Indications for surgery

  * Refractory retention (failed ≥1 trial of voiding).
  * Associated bladder Stones.
  * Associated recurrent gross Hematuria.
  * Associated with recurrent Infections.
  * Associated renal insufficiency.
  * Bother symptoms refractory to medical treatment.

Exclusion Criteria:

* Uncorrectable coagulopathy.
* Patient with active UTI.
* Prostate less than 80 ml.
* Severe associated comorbidities.
* Previous urethral, prostate, and bladder surgeries,
* Patients diagnosed with neurogenic bladder.
* Patients diagnosed with prostate cancer.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
operative time | Three months
  To measure the difference between the two procedure regarding operative time measured in minutes.
recovery outcome | Three months
  To measure the difference between the two procedure regarding mean hospital stays measured in days and catheterization period measured in days

SECONDARY OUTCOMES:
peri-operative complication | Three months
  to measure the difference between the two procedures regarding incidence of early complications including re-catheterization, acute urinary retention, early irritative symptoms and urinary tract infections and incidence of late complications Including urinary incontinence, Urethral strictures,and bladder neck contracture.
weight of resected prostatic tissues | Three months
  to measure the difference between the two procedures regarding weight of resected prostatic tissues Measured in gram
post-operative International Prostate Symptom Score (IPSS) score. | Three months
  to measure the difference between the two procedures regarding IPSS score. Score 0 to 7 points considered mild symptoms, 8 to 19 points considered moderate symptoms, 20 to 35 points considered severe symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Tarek Salem, professor, Study Director — Helwan university faculty of medicine
Locations (1):
- Helwan university faculty of medicine, Helwan, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mahon JT, McVary KT. New Alternative Treatments for Lower Urinary Tract Symptoms Secondary to Benign Prostatic Hyperplasia. Minimally Invasive Urology: Springer; 2020. p. 283-305.
- [Result] Barry MJ, Fowler FJ Jr, O'leary MP, Bruskewitz RC, Holtgrewe HL, Mebust WK, Cockett AT; Measurement Committee of the American Urological Association. The American Urological Association Symptom Index for Benign Prostatic Hyperplasia. J Urol. 2017 Feb;197(2S):S189-S197. doi: 10.1016/j.juro.2016.10.071. Epub 2016 Dec 22. PMID 28012747
- [Result] De Nunzio C, Lombardo R, Cicione AM, Tubaro A. Benign Prostatic Hyperplasia (BPH). Urologic Principles and Practice: Springer; 2020. p. 341-55.
- [Result] Foster HE, Barry MJ, Dahm P, Gandhi MC, Kaplan SA, Kohler TS, Lerner LB, Lightner DJ, Parsons JK, Roehrborn CG, Welliver C, Wilt TJ, McVary KT. Surgical Management of Lower Urinary Tract Symptoms Attributed to Benign Prostatic Hyperplasia: AUA Guideline. J Urol. 2018 Sep;200(3):612-619. doi: 10.1016/j.juro.2018.05.048. Epub 2018 Jun 11. PMID 29775639
- [Result] Zheng X, Han X, Cao D, Wang Y, Xu H, Yang L, Wei Q, Ai J. Comparison of Short-Term Outcomes between Button-Type Bipolar Plasma Vaporization and Transurethral Resection for the Prostate: A Systematic Review and Meta-Analysis. Int J Med Sci. 2019 Oct 21;16(12):1564-1572. doi: 10.7150/ijms.38618. eCollection 2019. PMID 31839744
- [Result] Xie L, Mao Q, Chen H, Qin J, Zheng X, Lin Y, Wang X, Liu B. Transurethral vapor enucleation and resection of the prostate with plasma vaporization button electrode for the treatment of benign prostatic hyperplasia: a feasibility study. J Endourol. 2012 Oct;26(10):1264-6. doi: 10.1089/end.2012.0125. Epub 2012 Sep 12. PMID 22530928
- [Result] Sagen E, Namnuan RO, Hedelin H, Nelzen O, Peeker R. The morbidity associated with a TURP procedure in routine clinical practice, as graded by the modified Clavien-Dindo system. Scand J Urol. 2019 Aug;53(4):240-245. doi: 10.1080/21681805.2019.1623312. Epub 2019 Jun 3. PMID 31156002
- [Result] Morton S, McGuiness L, Harding C, Thorpe A. A review of surgery and new technology procedures for the management of benign prostatic obstruction. Journal of Clinical Urology. 2019;12(6):474-86.
- [Result] Giulianelli R, Gentile BC, Mirabile G, Tema G, Albanesi L, Tariciotti P, Rizzo G, Falavolti C, Aloisi P, Vincenti G, Lombardo R. Bipolar plasma enucleation of the prostate vs. open prostatectomy in large benign prostatic hyperplasia: a single centre 3-year comparison. Prostate Cancer Prostatic Dis. 2019 Mar;22(1):110-116. doi: 10.1038/s41391-018-0080-7. Epub 2018 Aug 21. PMID 30131603
- [Result] Lokeshwar SD, Harper BT, Webb E, Jordan A, Dykes TA, Neal DE Jr, Terris MK, Klaassen Z. Epidemiology and treatment modalities for the management of benign prostatic hyperplasia. Transl Androl Urol. 2019 Oct;8(5):529-539. doi: 10.21037/tau.2019.10.01. PMID 31807429